CLINICAL TRIAL: NCT01421147
Title: A Prospective, Randomized, Open-label Comparison of a Long-Acting Basal Insulin Analog LY2963016 to Lantus in Combination With Mealtime Insulin Lispro in Adult Patients With Type 1 Diabetes Mellitus
Brief Title: A Study in Adults With Type 1 Diabetes
Acronym: ELEMENT 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13712; I4L-MC-ABEB (Other: Eli Lilly and Company); 2011-000829-73 (EudraCT Number)
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Type 1 Diabetes; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — LY2963016 insulin glargine; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2963016 + Insulin Lispro (Experimental): LY2963016 titrated based on blood glucose readings, administered subcutaneously, once daily at the same timing (daytime or evening/bedtime) as participant's prestudy basal insulin injection schedule in combination with premeal insulin lispro. Insulin lispro titrated based on blood glucose readings, administered subcutaneously, three times a day for 52 weeks.
  Interventions: Drug: LY2963016; Drug: Insulin Lispro
- Lantus + Insulin Lispro (Active Comparator): Lantus titrated based on blood glucose readings, administered subcutaneously, once daily at the same timing (daytime or evening/bedtime) as participant's prestudy basal insulin injection schedule in combination with premeal insulin lispro. Insulin lispro titrated based on blood glucose readings, administered subcutaneously, three times a day for 52 weeks.
  Interventions: Drug: Lantus; Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY2963016 — Administered subcutaneously
  Arms: LY2963016 + Insulin Lispro
Drug: Lantus — Administered subcutaneously
  Arms: Lantus + Insulin Lispro
Drug: Insulin Lispro — Administered subcutaneously

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of LY2963016 versus Lantus when taken once daily in combination with insulin lispro before meals three times a day.

ELIGIBILITY:
Inclusion Criteria:

* Have type 1 diabetes mellitus based on the disease diagnostic criteria [World Health Organization (WHO) Classification]
* Have duration of diabetes greater than or equal to one year
* Have Hemoglobin A1c (HbA1c) less than or equal to 11.0%
* On basal-bolus insulin therapy for at least 1 year [basal insulin must be once daily (QD) injection of human insulin isophane suspension (NPH), Lantus, or detemir and combined with mealtime injections of human regular insulin, or insulin analog lispro, aspart or glulisine]
* Have a body mass index (BMI) of less than or equal to 35 kilograms/square meter (kg/m²)

Exclusion Criteria:

* Have had more than one episode of severe low blood sugar (defined as needing someone else to help because you had very low blood sugar) within the 6 months before entering the study
* Have had more than one episode of diabetic ketoacidosis or emergency room visits for uncontrolled diabetes leading to hospitalization within the 6 months before entering the study
* Have known hypersensitivity or allergy to any of the study insulins (insulin glargine or insulin lispro) or to excipients of the study insulins
* Have significant renal, cardiac, gastrointestinal or liver disease
* Have active cancer or cancer within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (52):
- United States (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roswell, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mineola, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Hyde Park, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., LiÃ¨ge
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fulda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Ingbert-OberwÃ¼rzbach
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haidari/Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salgótarján
- Japan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyazaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Puebla City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
- Romania (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara

REFERENCES:
- [Derived] Nishiyama H, Shingaki T, Suzuki Y, Ilag LL. Similar Intrapatient Blood Glucose Variability with LY2963016 and Lantus(R) Insulin Glargine in Patients with Type 1 (T1D) or Type 2 Diabetes, Including a Japanese T1D Subpopulation. Diabetes Ther. 2018 Aug;9(4):1469-1476. doi: 10.1007/s13300-018-0450-0. Epub 2018 May 31. PMID 29855972

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 24-week treatment period followed by a 28-week extension period.
Groups:
- LY2963016 + Insulin Lispro: LY2963016 dose was titrated based on blood glucose readings, and administered subcutaneously, once daily at the same timing (daytime or evening/bedtime) as participant's prestudy basal insulin injection schedule in combination with premeal insulin lispro for 52 weeks. Insulin lispro dosing was titrated based on blood glucose readings, and administered subcutaneously, 3 times a day for 52 weeks.
- Lantus + Insulin Lispro: Lantus dose was titrated based on blood glucose readings, and administered subcutaneously, once daily at the same timing (daytime or evening/bedtime) as participant's prestudy basal insulin injection schedule in combination with premeal insulin lispro for 52 weeks. Insulin lispro dosing was titrated based on blood glucose readings, and administered subcutaneously, 3 times a day for 52 weeks.
Period: Treatment Period
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Started | 269 | 267
Received at Least 1 Dose of Study Drug | 268 | 267
Completed | 253 | 256
Not Completed | 16 | 11
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 10 | 5
Period: Extension Period
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Started | 253 | 256
Completed | 245 | 245
Not Completed | 8 | 11
Not completed — Adverse Event | 0 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro | Total
Number analyzed (Participants) | 268 | 267 | 535
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.96 (13.65) | 41.37 (13.25) | 41.16 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 112 | 225
  Male | 155 | 155 | 310
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 21
  Not Hispanic or Latino | 177 | 170 | 347
  Unknown or Not Reported | 80 | 87 | 167
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 12 | 23
  Asian | 49 | 51 | 100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 2 | 11
  White | 197 | 201 | 398
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 99 | 96 | 195
  Hungary | 14 | 16 | 30
  Mexico | 17 | 19 | 36
  Greece | 15 | 13 | 28
  Belgium | 12 | 11 | 23
  Poland | 18 | 17 | 35
  Romania | 18 | 16 | 34
  Germany | 26 | 28 | 54
  Japan | 49 | 51 | 100
Baseline Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — HbA1c is the glycosylated fraction of hemoglobin A which provides an estimate of a participant's blood sugar control over a 6- to 12-week period.
  percentage of glycosylated hemoglobin | 7.75 (1.13) | 7.79 (1.03) | 7.77 (1.08)
Time of Basal Insulin Injection [Number; unit: participants] — Number of participants who administered a basal insulin injection during the Daytime and Evening/Bedtime.
  participants
    Daytime | 51 | 48 | 99
    Evening/Bedtime | 217 | 219 | 436
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 75.80 (16.76) | 74.77 (15.36) | 75.29 (16.07)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline up to 24 Weeks in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A which provides an estimate of a participant's blood sugar control over a 6- to 12-week period. Least Squares (LS) means were calculated by analysis of covariance (ANCOVA) and adjusted for baseline HbA1c, treatment and time of basal insulin injection (daytime, evening/bedtime) and country.
Time Frame: Baseline, Endpoint (up to 24 weeks)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline HbA1c measurement. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 267 | 267
percentage of glycosylated hemoglobin | -0.352 (0.053) | -0.460 (0.054)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.055, ANCOVA; LS Mean Difference = 0.108, 95% CI 2-sided [-0.002 to 0.219]

2. Secondary Outcome: Change From Baseline in Insulin Antibody Levels
Description: Blood samples are collected from participants and percentage of insulin antibody binding was measured to determine the insulin antibody levels. Least Squares (LS) means were calculated by analysis of covariance (ANCOVA) and adjusted for baseline hemoglobin A1c (HbA1c), treatment and time of basal insulin injection (daytime, evening/bedtime) and country.
Time Frame: Baseline, 6 weeks and 12 weeks and Endpoints (up to 24 weeks and up to 52 weeks)
Population: All randomized participants who received at least 1 dose of study drug and were insulin antibody positive at baseline and had at least 1 post-baseline insulin antibody positive measurement. Last observation carried forward (LOCF) principle was used for Endpoints (up to 24 and up to 52 weeks).
Measure: Least Squares Mean (Standard Error); unit: percentage of insulin antibody binding
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 40 | 47
percentage of insulin antibody binding
  Change at 6 weeks (n=31, 38) | 0.30 (0.33) | -0.12 (0.33)
  Change at 12 weeks (n=27, 36) | 0.02 (0.39) | -0.38 (0.39)
  Change at Endpoint, up to 24 weeks (n=37, 47) | 0.47 (0.45) | 0.09 (0.44)
  Change at Endpoint, up to 52 weeks (n=40, 47) | 0.87 (0.58) | 0.06 (0.56)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.205, ANCOVA — P-value is for change at 6 weeks; LS Mean Difference = 0.41, 95% CI 2-sided [-0.23 to 1.05]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.320, ANCOVA — P-value is for change at 12 weeks; LS Mean difference = 0.40, 95% CI 2-sided [-0.40 to 1.21]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.373, ANCOVA — P-value is for change at Endpoint, up to 24 weeks; LS Mean Difference = 0.37, 95% CI 2-sided [-0.46 to 1.21]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.131, ANCOVA — P-value is for change at Endpoint, up to 52 weeks; LS Mean Difference = 0.81, 95% CI 2-sided [-0.25 to 1.86]

3. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: as for outcome 1
Time Frame: Baseline, 6 weeks and 12 weeks and 24 weeks and 36 weeks and 52 weeks and Endpoint (up to 52 weeks)
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline HbA1c measurements. Last observation carried forward (LOCF) principle was used for Endpoint (up to 52 weeks).
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 267 | 267
percentage of glycosylated hemoglobin
  Change at 6 weeks (n=265, 265) | -0.369 (0.038) | -0.362 (0.039)
  Change at 12 weeks (n=261, 262) | -0.359 (0.049) | -0.472 (0.049)
  Change at 24 weeks (n=256, 258) | -0.383 (0.053) | -0.481 (0.053)
  Change at 36 weeks (n=253, 254) | -0.349 (0.056) | -0.408 (0.056)
  Change at 52 weeks (n=248, 246) | -0.302 (0.059) | -0.306 (0.060)
  Change at Endpoint, up to 52 weeks (n=267, 267) | -0.256 (0.057) | -0.276 (0.058)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.860, ANCOVA — P-value is for change at 6 weeks; LS Mean Difference = -0.007, 95% CI 2-sided [-0.087 to 0.072]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.030, ANCOVA — P-value is for change at 12 weeks; LS Mean Difference = 0.113, 95% CI 2-sided [0.011 to 0.215]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.080, ANCOVA — P-value is for change at 24 weeks; LS Mean Difference = 0.098, 95% CI 2-sided [-0.012 to 0.208]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.314, ANCOVA — P-value is for change at 36 weeks; LS Mean Difference = 0.060, 95% CI 2-sided [-0.057 to 0.177]
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.948, ANCOVA — P-value is for change at 52 weeks; LS Mean Difference = 0.004, 95% CI 2-sided [-0.119 to 0.127]
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.737, ANCOVA — P-value is for change at Endpoint, up to 52 weeks; LS Mean Difference = 0.020, 95% CI 2-sided [-0.099 to 0.140]

4. Secondary Outcome: 7-Point Self-Monitored Blood Glucose (SMBG) Profiles
Description: 7-point SMBG measurements are completed at the following timepoints: Morning (AM) Pre-Meal, AM Post-Prandial (PP), Midday (MD) Pre-Meal, MD PP, Evening (EV) Pre-Meal, Bed Time and 0300 hours. PP glucose is measured 2 hours (hrs) after the start of the meal. Values for the 7-point SMBG profiles were averaged over the three 7-point SMBG profiles during 2-week period prior to each visit. If only 1 of the 3 days of data was collected, then the value of the 1 day was used. If only 2 of the 3 days of data were collected, then the average of the 2 days was used. Least Squares (LS) means were calculated by analysis of covariance (ANCOVA) and adjusted for baseline hemoglobin A1c (HbA1c), treatment and time of basal insulin injection (daytime, evening/bedtime) and country.
Time Frame: Baseline and Endpoints [up to 24 weeks (wk) and up to 52 weeks]
Population: All randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline SMBG measurement. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 266 | 265
millimoles per liter (mmol/L)
  Baseline-AM Pre-Meal (n=266, 264) | 8.37 (0.18) | 8.19 (0.18)
  Baseline-AM 2 hrs PP (n=263, 262) | 8.93 (0.19) | 9.41 (0.19)
  Baseline-MD Pre-Meal (n=266, 265) | 7.86 (0.16) | 8.14 (0.16)
  Baseline-MD 2 hrs PP (n=264, 264) | 9.12 (0.18) | 8.81 (0.18)
  Baseline-EV Pre-Meal (n=264, 264) | 8.87 (0.19) | 8.82 (0.19)
  Baseline-Bed Time (n=266, 264) | 9.26 (0.20) | 9.37 (0.20)
  Baseline-0300 hrs (n=262, 257) | 8.27 (0.18) | 8.37 (0.18)
  Endpoint, up to 24 wk-AM Pre-Meal (n=266, 264) | 7.98 (0.20) | 7.81 (0.20)
  Endpoint, up to 24 wk-AM 2 hrs PP (n=263, 262) | 8.75 (0.20) | 8.50 (0.21)
  Endpoint, up to 24 wk-MD Pre-Meal (n=266, 265) | 7.81 (0.19) | 7.84 (0.20)
  Endpoint, up to 24 wk-MD 2 hrs PP (n=264, 264) | 8.50 (0.21) | 8.41 (0.21)
  Endpoint, up to 24 wk-EV Pre-Meal (n=264, 264) | 8.82 (0.21) | 8.61 (0.22)
  Endpoint, up to 24 wk-Bed Time (n=266, 264) | 8.61 (0.22) | 9.11 (0.22)
  Endpoint, up to 24 wk-0300 hrs (n=262, 257) | 7.93 (0.20) | 8.38 (0.20)
  Endpoint, up to 52 wk- AM Pre-Meal (n=266, 264) | 8.03 (0.20) | 8.29 (0.21)
  Endpoint, up to 52 wk-AM 2 hrs PP (n=263, 262) | 8.55 (0.21) | 8.88 (0.21)
  Endpoint, up to 52 wk-MD Pre-Meal (n=266, 265) | 7.96 (0.19) | 7.99 (0.19)
  Endpoint, up to 52 wk-MD 2 hrs PP (n=264, 264) | 8.61 (0.21) | 8.74 (0.21)
  Endpoint, up to 52 wk-EV Pre-Meal (n=264, 264) | 8.37 (0.21) | 8.38 (0.21)
  Endpoint, up to 52 wk-Bed Time (n=266, 264) | 8.57 (0.21) | 9.06 (0.21)
  Endpoint, up to 52 wk-0300 hrs (n=262, 257) | 8.22 (0.21) | 8.43 (0.22)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.489, ANCOVA — P-value is for Baseline-AM Pre-Meal; LS Mean Difference = 0.18, 95% CI 2-sided [-0.33 to 0.69]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.066, ANCOVA — P-value is for Baseline-AM 2 hrs PP; LS Mean Difference = -0.48, 95% CI 2-sided [-1.00 to 0.03]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.209, ANCOVA — P-value is for Baseline-MD Pre-Meal; LS Mean Difference = -0.28, 95% CI 2-sided [-0.71 to 0.16]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.232, ANCOVA — P-value is for Baseline-MD 2 hrs PP; LS Mean Difference = 0.31, 95% CI 2-sided [-0.20 to 0.82]
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.856, ANCOVA — P-value is for Baseline-EV Pre-Meal; LS Mean Difference = 0.05, 95% CI 2-sided [-0.49 to 0.58]
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.693, ANCOVA — P-value is for Baseline-Bed Time; LS Mean Difference = -0.11, 95% CI 2-sided [-0.66 to 0.44]
Statistical Analysis 7: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.700, ANCOVA — P-value is for Baseline-0300 hrs; LS Mean Difference = -0.10, 95% CI 2-sided [-0.61 to 0.41]
Statistical Analysis 8: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.399, ANCOVA — P-value is for Endpoint, up to 24 wk-AM Pre-Meal; LS Mean Difference = 0.17, 95% CI 2-sided [-0.23 to 0.58]
Statistical Analysis 9: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.248, ANCOVA — P-value is for Endpoint, up to 24 wk-AM 2 hrs PP; LS Mean Difference = 0.25, 95% CI 2-sided [-0.18 to 0.68]
Statistical Analysis 10: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.883, ANCOVA — P-value is for Endpoint, up to 24 wk-MD Pre-Meal; LS Mean Difference = -0.03, 95% CI 2-sided [-0.44 to 0.38]
Statistical Analysis 11: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.687, ANCOVA — P-value is for Endpoint, up to 24 wk-MD 2 hrs PP; LS Mean Difference = 0.09, 95% CI 2-sided [-0.34 to 0.52]
Statistical Analysis 12: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.364, ANCOVA — P-value is for Endpoint, up to 24 wk-EV Pre-Meal; LS Mean Difference = 0.20, 95% CI 2-sided [-0.24 to 0.65]
Statistical Analysis 13: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.030, ANCOVA — P-value is for Endpoint, up to 24 wk- Bed Time; LS Mean Difference = -0.50, 95% CI 2-sided [-0.95 to -0.05]
Statistical Analysis 14: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.033, ANCOVA — P-value is for Endpoint, up to 24 wk-0300 hrs; LS Mean Difference = -0.45, 95% CI 2-sided [-0.86 to -0.04]
Statistical Analysis 15: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.230, ANCOVA — P-value is for Endpoint, up to 52 wk-AM Pre-Meal; LS Mean Difference = -0.26, 95% CI 2-sided [-0.68 to 0.16]
Statistical Analysis 16: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.148, ANCOVA — P-value is for Endpoint, up to 52 wk-AM 2 hrs PP; LS Mean Difference = -0.32, 95% CI 2-sided [-0.76 to 0.11]
Statistical Analysis 17: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.866, ANCOVA — P-value is for Endpoint, up to 52 wk-MD Pre-Meal; LS Mean Difference = -0.03, 95% CI 2-sided [-0.43 to 0.36]
Statistical Analysis 18: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.545, ANCOVA — P-value is for Endpoint, up to 52 wk-MD 2 hrs PP; LS Mean Difference = -0.13, 95% CI 2-sided [-0.56 to 0.30]
Statistical Analysis 19: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.955, ANCOVA — P-value is for Endpoint, up to 52 wk-EV Pre-Meal; LS Mean Difference = -0.01, 95% CI 2-sided [-0.44 to 0.42]
Statistical Analysis 20: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.031, ANCOVA — P-value is for Endpoint, up to 52 wk-Bed Time; LS Mean Difference = -0.48, 95% CI 2-sided [-0.92 to -0.04]
Statistical Analysis 21: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.355, ANCOVA — P-vale is for Endpoint, up to 52 wk-0300 hrs; LS Mean Difference = -0.21, 95% CI 2-sided [-0.65 to 0.23]

5. Secondary Outcome: Glycemic Variability of Fasting Blood Glucose
Description: Glycemic variability is the intra-participant standard deviation (SD) value of fasting blood glucose as measured by the actual morning premeal blood glucose value from the 7-point self-monitoring blood glucose (SMBG) profiles. Least Squares (LS) means were calculated by analysis of covariance (ANCOVA) and adjusted for baseline hemoglobin A1c (HbA1c), treatment and time of basal insulin injection (daytime, evening/bedtime) and country.
Time Frame: Baseline and Endpoints (up to 24 weeks and up 52 weeks)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline fasting blood glucose measurement. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 264 | 259
millimoles per liter (mmol/L)
  Baseline | 2.51 (0.12) | 2.68 (0.12)
  Endpoint, up to 24 weeks | 2.25 (0.14) | 2.29 (0.14)
  Endpoint, up to 52 weeks | 2.08 (0.13) | 2.34 (0.13)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.320, ANCOVA — P-value is for Baseline; LS Mean Difference = -0.17, 95% CI 2-sided [-0.52 to 0.17]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.781, ANCOVA — P-value is for Endpoint, up to 24 weeks; LS Mean Difference = -0.04, 95% CI 2-sided [-0.33 to 0.25]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.060, ANCOVA — P-value is for Endpoint, up to 52 weeks; LS Mean Difference = -0.26, 95% CI 2-sided [-0.53 to 0.01]

6. Secondary Outcome: Change From Baseline in Body Weight
Description: Least Squares (LS) means were calculated by analysis of covariance (ANCOVA) and adjusted for baseline hemoglobin A1c (HbA1c), treatment and time of basal insulin injection (daytime, evening/bedtime) and country.
Time Frame: Baseline, 6 weeks and 12 weeks and 18 weeks and Endpoints (up to 24 weeks and up to 52 weeks)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline body weight measurement. Last observation carried forward (LOCF) principle was used for Endpoints (up to 24 weeks and up to 52 weeks).
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 268 | 267
kilogram (kg)
  Change at 6 weeks (n=265, 265) | 0.45 (0.09) | 0.42 (0.09)
  Change at 12 weeks (n=261, 261) | 0.59 (0.13) | 0.48 (0.13)
  Change at 18 weeks (n=258, 260) | 0.72 (0.15) | 0.55 (0.15)
  Change at Endpoint, up to 24 weeks (n=268, 267) | 0.66 (0.17) | 0.42 (0.17)
  Change at Endpoint, up to 52 weeks (n=268, 267) | 0.93 (0.21) | 0.59 (0.21)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.823, ANCOVA — P-value is for change at 6 weeks; LS Mean Difference = 0.03, 95% CI 2-sided [-0.23 to 0.29]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.541, ANCOVA — P-value is for change at 12 weeks; LS Mean Difference = 0.11, 95% CI 2-sided [-0.25 to 0.47]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.435, ANCOVA — P-value is for change at 18 weeks; LS Mean Difference = 0.17, 95% CI 2-sided [-0.25 to 0.59]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.320, ANCOVA — P-value is for change at Endpoint, up to 24 weeks; LS Mean Difference = 0.24, 95% CI 2-sided [-0.23 to 0.71]
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.253, ANCOVA — P-value is for change at Endpoint, up to 52 weeks; LS Mean Difference = 0.34, 95% CI 2-sided [-0.25 to 0.93]

7. Secondary Outcome: Adult Low Blood Sugar Survey (ALBSS)
Description: ALBSS contains 33 items, with each item scored on a 5-point response scale: 0 (never) to 4 (almost always). Items are categorized in 2 domains: Behavior (or avoidance) Items 1 to 15 and Worry (or affect) Items 16 to 33. Behavior Total Score (TS) range is 0 to 60 and Worry TS range is 0 to 72. Higher scores on "Behavior" items (related to avoidance of hypoglycemia) reflect greater awareness and/or effort of the participant to prevent low blood sugar. Higher scores on "Worry" items (related to worries about low blood sugar and its consequences) reflect greater participant concern about having low blood sugar. Least Squares (LS) means were calculated by analysis of covariance (ANCOVA) and adjusted for baseline hemoglobin A1c (HbA1c), treatment and time of basal insulin injection (daytime, evening/bedtime) and country.
Time Frame: Baseline and 24 weeks and Endpoint (up to 52 weeks)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline ALBSS measurement. Last observation carried forward (LOCF) principle was used for Endpoint (up to 52 weeks).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 265 | 263
units on a scale
  Baseline-Behavior TS (n=265, 263) | 13.63 (0.54) | 12.99 (0.54)
  24 weeks-Behavior TS (n=255, 257) | 12.73 (0.66) | 12.53 (0.66)
  Endpoint, up to 52 weeks-Behavior TS (n=265, 263) | 13.19 (0.62) | 13.03 (0.62)
  Baseline-Worry TS (n=265, 263) | 16.01 (0.83) | 14.81 (0.83)
  24 weeks-Worry TS (n=255, 258) | 15.39 (1.08) | 14.27 (1.08)
  Endpoint, up to 52 weeks-Worry TS (n=265, 263) | 15.18 (1.03) | 14.93 (1.05)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.401, ANCOVA — P-value is for Baseline-Behavior TS; LS Mean Difference = 0.64, 95% CI 2-sided [-0.86 to 2.15]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.778, ANCOVA — P-value is for 24 weeks-Behavior TS; LS Mean Difference = 0.20, 95% CI 2-sided [-1.16 to 1.55]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.804, ANCOVA — P-value is for Endpoint, up to 52 weeks-Behavior TS; LS Mean Difference = 0.16, 95% CI 2-sided [-1.12 to 1.45]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.304, ANCOVA — P-value is for Baseline-Worry TS; LS Mean Difference = 1.21, 95% CI [-1.10 to 3.51]
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.323, ANCOVA — P-value is for 24 weeks-Worry TS; LS Mean Difference = 1.12, 95% CI 2-sided [-1.10 to 3.34]
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.824, ANCOVA — P-value is for Endpoint, up to 52 weeks-Worry TS; LS Mean Difference = 0.25, 95% CI [-1.92 to 2.41]

8. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ)
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. Items measured on a 7-point scale: 1 (no bother at all) to 7 (a tremendous bother), with lower scores reflecting better outcomes. Items divided into 5 domains: Inconvenience of Regimen [(IR) 5 items: scores range 5-35], Lifestyle Flexibility [(LF) 3 items: scores range 3-21], Glycemic Control [(GC) 3 items: scores range 3-21], Hypoglycemic Control [(HC) 5 items: scores range 5-35], Insulin Delivery Device [(IDD) 6 items: scores range 6-42]. ITSQ Total Overall Scores range from 22-154. Data presented are the transformed score on a scale of 0-100, where transformed score=100×[(7-raw score)/6]. Higher scores indicate better treatment satisfaction. Least Squares (LS) means were calculated by analysis of covariance (ANCOVA) and adjusted for baseline hemoglobin A1c (HbA1c), treatment and time of basal insulin injection (daytime, evening/bedtime) and country.
Time Frame: Baseline and 24 weeks and Endpoint (up to 52 weeks)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline ITSQ measurements. Last observation carried forward (LOCF) principle was used for Endpoint (up to 52 weeks).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 264 | 262
units on a scale
  IR-Baseline (n=264, 263) | 74.62 (1.31) | 75.39 (1.32)
  IR-24 weeks (n=254, 258) | 79.32 (1.62) | 78.76 (1.62)
  IR-Endpoint, up to 52 weeks (n=264, 263) | 79.50 (1.60) | 80.44 (1.62)
  LF-Baseline (n=264, 263) | 63.19 (1.47) | 62.38 (1.47)
  LF-24 weeks (n=254, 258) | 64.18 (1.90) | 63.34 (1.90)
  LF-Endpoint, up to 52 weeks (n=264, 263) | 63.25 (1.86) | 64.16 (1.88)
  GC-Baseline (n=264, 263) | 64.44 (1.34) | 64.34 (1.34)
  GC-24 weeks (n=254, 258) | 72.99 (1.62) | 71.73 (1.62)
  GC-Endpoint, up to 52 weeks (n=264, 263) | 70.15 (1.67) | 69.24 (1.69)
  HC-Baseline (n=264, 263) | 70.20 (1.15) | 70.81 (1.15)
  HC-24 weeks (n=254, 258) | 70.40 (1.48) | 71.42 (1.48)
  HC-Endpoint, up to 52 weeks (n=264, 263) | 70.46 (1.47) | 71.72 (1.49)
  IDD-Baseline (n=262, 262) | 75.22 (1.20) | 76.75 (1.20)
  IDD-24 weeks (n=252, 258) | 79.77 (1.42) | 79.36 (1.42)
  IDD-Endpoint, up to 52 weeks (n=262, 262) | 79.46 (1.37) | 79.75 (1.39)
  ITSQ Total-Baseline (n=264, 262) | 70.80 (0.99) | 71.39 (1.00)
  ITSQ Total-24 weeks (n=253, 258) | 74.46 (1.23) | 74.23 (1.24)
  ITSQ Total-Endpoint, up to 52 weeks (n=264, 262) | 73.94 (1.25) | 74.48 (1.26)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.681, ANCOVA — P-value is for IR-Baseline; LS Mean Difference = -0.77, 95% CI 2-sided [-4.42 to 2.89]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.744, ANCOVA — P-value is for IR-24 weeks; LS Mean Difference = 0.56, 95% CI 2-sided [-2.79 to 3.90]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.582, ANCOVA — P-value is for IR-Endpoint, up to 52 weeks; LS Mean Difference = -0.94, 95% CI 2-sided [-4.29 to 2.41]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.694, ANCOVA — P-value is for LF-Baseline; LS Mean Difference = 0.82, 95% CI 2-sided [-3.26 to 4.89]
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.673, ANCOVA — P-value is for LF-24 weeks; LS Mean Difference = 0.84, 95% CI 2-sided [-3.08 to 4.77]
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.645, ANCOVA — P-value is for LF-Endpoint, up to 52 weeks; LS Mean Difference = -0.91, 95% CI 2-sided [-4.79 to 2.97]
Statistical Analysis 7: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.961, ANCOVA — P-value is for GC-Baseline; LS Mean Difference = 0.09, 95% CI 2-sided [-3.62 to 3.81]
Statistical Analysis 8: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.463, ANCOVA — P-value is for GC-24 weeks; LS Mean Difference = 1.25, 95% CI 2-sided [-2.10 to 4.61]
Statistical Analysis 9: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.609, ANCOVA — P-value is for GC-Endpoint, up to 52 weeks; LS Mean Difference = 0.91, 95% CI 2-sided [-2.59 to 4.41]
Statistical Analysis 10: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.708, ANCOVA — P-value is for HC-Baseline; LS Mean Difference = -0.61, 95% CI 2-sided [-3.81 to 2.59]
Statistical Analysis 11: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.510, ANCOVA — P-value is for HC-24 weeks; LS Mean Difference = -1.03, 95% CI 2-sided [-4.09 to 2.03]
Statistical Analysis 12: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.422, ANCOVA — P-value is for HC-Endpoint, up to 52 weeks; LS Mean Difference = -1.26, 95% CI 2-sided [-4.34 to 1.82]
Statistical Analysis 13: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.367, ANCOVA — P-value is for IDD-Baseline; LS Mean Difference = -1.53, 95% CI 2-sided [-4.85 to 1.80]
Statistical Analysis 14: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.786, ANCOVA — P-value is for IDD-24 weeks; LS Mean Difference = 0.41, 95% CI 2-sided [-2.54 to 3.35]
Statistical Analysis 15: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.845, ANCOVA — P-value is for IDD-Endpoint, up to 52 weeks; LS Mean Difference = -0.29, 95% CI 2-sided [-3.16 to 2.59]
Statistical Analysis 16: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.676, ANCOVA — P-value is for ITSQ Total-Baseline; LS Mean Difference = -0.59, 95% CI 2-sided [-3.36 to 2.18]
Statistical Analysis 17: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.862, ANCOVA — P-value is for ITSQ Total-24 weeks; LS Mean Difference = 0.23, 95% CI 2-sided [-2.33 to 2.78]
Statistical Analysis 18: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.685, ANCOVA — P-value is for ITSQ Total-Endpoint, up to 52 weeks; LS Mean Difference = -0.54, 95% CI 2-sided [-3.15 to 2.07]

9. Secondary Outcome: Insulin Dose Per Body Weight (U/kg) (Total and by Component [Basal and Bolus (Lispro)])
Description: Total daily insulin dose was adjusted for body weight [units of insulin/kilogram/day (U/kg/day)]. Least Squares (LS) means were calculated by analysis of covariance (ANCOVA) and adjusted for baseline hemoglobin A1c (HbA1c), treatment and time of basal insulin injection (daytime, evening/bedtime) and country.
Time Frame: Endpoints [up to 24 weeks (wk) and up to 52 weeks]
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 daily insulin dose per body weight measurements. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: U/kg/day
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 268 | 266
U/kg/day
  Endpoint, up to 24 wk-Basal Insulin (n=268, 266) | 0.371 (0.011) | 0.358 (0.011)
  Endpoint, up to 24 wk-Bolus Insulin (n=264, 266) | 0.352 (0.015) | 0.346 (0.016)
  Endpoint, up to 24 wk-Total Insulin (n=264, 266) | 0.723 (0.021) | 0.704 (0.021)
  Endpoint, up to 52 wk-Basal Insulin (n=268, 266) | 0.379 (0.012) | 0.361 (0.012)
  Endpoint, up to 52 wk-Bolus Insulin (n=264, 266) | 0.369 (0.016) | 0.370 (0.016)
  Endpoint, up to 52 wk-Total Insulin (n=264, 266) | 0.748 (0.022) | 0.731 (0.022)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.235, ANCOVA — P-value is for Endpoint, up to 24 wk-Basal Insulin; LS Mean Difference = 0.014, 95% CI 2-sided [-0.009 to 0.036]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.726, ANCOVA — P-value is for Endpoint, up to 24 wk-Bolus Insulin; LS Mean Difference = 0.006, 95% CI 2-sided [-0.026 to 0.038]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.377, ANCOVA — P-value is for Endpoint, up to 24 wk-Total Insulin; LS Mean Difference = 0.019, 95% CI 2-sided [-0.023 to 0.062]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.159, ANCOVA — P-value is for Endpoint, up to 52 wk-Basal Insulin; LS Mean Difference = 0.018, 95% CI 2-sided [-0.007 to 0.042]
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.957, ANCOVA — P-value is for Endpoint, up to 52 wk-Bolus Insulin; LS Mean Difference = -0.001, 95% CI 2-sided [-0.034 to 0.032]
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.450, ANCOVA — P-value is for Endpoint, up to 52 wk-Total Insulin; LS Mean Difference = 0.017, 95% CI 2-sided [-0.028 to 0.062]

10. Secondary Outcome: Insulin Dose - Units [Total and by Component [Basal and Bolus (Lispro)])
Description: Units of insulin taken daily were presented. Least Squares (LS) means were calculated by analysis of covariance (ANCOVA) and adjusted for baseline hemoglobin A1c (HbA1c), treatment and time of basal insulin injection (daytime, evening/bedtime) and country.
Time Frame: Endpoints [up to 24 weeks (wk) and up to 52 weeks]
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 insulin daily dose measurements. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: units of insulin per day (U/day)
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 268 | 266
units of insulin per day (U/day)
  Endpoint, up to 24 wk-Basal Insulin (n=268, 266) | 27.773 (0.970) | 26.049 (0.987)
  Endpoint, up to 24 wk-Bolus Insulin (n=264, 266) | 26.337 (1.347) | 25.069 (1.362)
  Endpoint, up to 24 wk-Total Insulin (n=264, 266) | 54.118 (1.948) | 51.154 (1.970)
  Endpoint, up to 52 wk-Basal Insulin (n=268, 266) | 28.463 (1.073) | 26.404 (1.091)
  Endpoint, up to 52 wk-Bolus Insulin (n=264, 266) | 27.800 (1.329) | 27.098 (1.344)
  Endpoint, up to 52 wk-Total Insulin (n=264, 266) | 56.255 (2.008) | 53.454 (2.031)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.096, ANCOVA — P-value is for Endpoint, up to 24 wk-Basal Insulin; LS Mean Difference = 1.724, 95% CI 2-sided [-0.308 to 3.755]
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.374, ANCOVA — P-value is for Endpoint, up to 24 wk-Bolus Insulin; LS Mean Difference = 1.267, 95% CI 2-sided [-1.531 to 4.065]
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.151, ANCOVA — P-value is for Endpoint, up to 24 wk-Total Insulin; LS Mean Difference = 2.964, 95% CI 2-sided [-1.081 to 7.010]
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.072, ANCOVA — P-value is for Endpoint, up to 52 wk-Basal Insulin; LS Mean Difference = 2.059, 95% CI 2-sided [-0.187 to 4.305]
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.617, ANCOVA — P-value is for Endpoint, up to 52 wk-Bolus Insulin; LS Mean Difference = 0.702, 95% CI 2-sided [-2.058 to 3.462]
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.188, ANCOVA — P-value is for Endpoint, up to 52 wk-Total Insulin; LS Mean Difference = 2.800, 95% CI 2-sided [-1.370 to 6.971]

11. Secondary Outcome: Percentage of Participants With Hemoglobin A1c (HbA1c) <7.0% and HbA1c ≤6.5%
Description: HbA1c is the glycosylated fraction of hemoglobin A which provides an estimate of a participant's blood sugar control over a 6- to 12-week period. The percentage of participants with Hemoglobin A1c (HbA1c) <7.0% or HbA1c ≤6.5% is calculated as the number of participants with an HbA1c level of the cut-off value (<7.0% or ≤6.5%) divided by the number of participants treated, then multiplied by 100.
Time Frame: Baseline and 6 weeks and 12 weeks and 24 weeks and 36 weeks and 52 weeks and Endpoints (up to 24 weeks and up to 52 weeks)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline HbA1c measurement. Last observation carried forward (LOCF) principle was used for Endpoints (up to 24 weeks and up to 52 weeks).
Measure: Number; unit: percentage of participants
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 267 | 267
percentage of participants
  HbA1c- at Baseline <7.0 % (n=267, 267) | 28.8 | 19.5
  HbA1c- at Baseline ≤6.5% (n=267, 267) | 13.9 | 12.0
  HbA1c- at 6 weeks <7.0% (n=265, 265) | 37.0 | 26.4
  HbA1c- at 6 weeks ≤6.5% (n=265, 265) | 21.1 | 14.3
  HbA1c- at 12 weeks <7.0% (n=261, 262) | 33.3 | 29.8
  HbA1c- at 12 weeks ≤6.5% (n=261, 262) | 19.9 | 15.3
  HbA1c- at 24 weeks <7.0% (n=256, 258) | 34.0 | 33.3
  HbA1c- at 24 weeks ≤6.5% (n=256, 258) | 19.9 | 19.0
  HbA1c- at 36 weeks <7.0% (n=253, 254) | 32.0 | 28.3
  HbA1c- at 36 weeks ≤6.5% (n=253, 254) | 15.4 | 18.5
  HbA1c- at 52 weeks <7.0% (n=248, 246) | 29.8 | 27.2
  HbA1c- at 52 weeks ≤6.5% (n=248, 246) | 15.3 | 14.6
  HbA1c- Endpoint, up to 24 weeks <7.0% (n=267, 267) | 34.5 | 32.2
  HbA1c- Endpoint, up to 24 weeks ≤6.5% (n=267, 267) | 20.2 | 18.4
  HbA1c- Endpoint, up to 52 weeks <7.0% (n=267, 267) | 30.3 | 25.1
  HbA1c- Endpoint, up to 52 weeks ≤6.5% (n=267, 267) | 15.7 | 13.5
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.015, Fisher Exact — P-value is for HbA1c- at Baseline <7.0 %
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.606, Fisher Exact — P-value is for HbA1c- at Baseline ≤6.5%
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.012, Fisher Exact — P-value is for HbA1c- at 6 weeks <7.0%
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.053, Fisher Exact — P-value is for HbA1c- at 6 weeks ≤6.5%
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.398, Fisher Exact — P-value is for HbA1c- at 12 weeks <7.0%
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.170, Fisher Exact — P-value is for HbA1c- at 12 weeks ≤6.5%
Statistical Analysis 7: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.926, Fisher Exact — P-value is for HbA1c- at 24 weeks <7.0%
Statistical Analysis 8: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.824, Fisher Exact — P-value is for HbA1c- at 24 weeks ≤6.5%
Statistical Analysis 9: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.385, Fisher Exact — P-value is for HbA1c- at 36 weeks <7.0%
Statistical Analysis 10: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.408, Fisher Exact — P-value is for HbA1c- at 36 weeks ≤6.5%
Statistical Analysis 11: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.551, Fisher Exact — P-value is for HbA1c- at 52 weeks <7.0%
Statistical Analysis 12: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.900, Fisher Exact — P-value is for HbA1c- at 52 weeks ≤6.5%
Statistical Analysis 13: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.646, Fisher Exact — P-value is for HbA1c- Endpoint, up to 24 weeks <7.0%
Statistical Analysis 14: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.661, Fisher Exact — P-value is for HbA1c- Endpoint, up to 24 weeks ≤6.5%
Statistical Analysis 15: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.209, Fisher Exact — P-value is for HbA1c- Endpoint, up to 52 weeks <7.0%
Statistical Analysis 16: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.540, Fisher Exact — P-value is for HbA1c- Endpoint, up to 52 weeks ≤6.5%

12. Secondary Outcome: Incidence of Hypoglycemic Events
Description: Incidence of hypoglycemic events is defined as the number of hypoglycemic events. A hypoglycemic event is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia, or has a blood glucose (BG) concentration of ≤ 70 milligrams/deciliter [mg/dL (3.9 millimoles/liter (mmol/L)], even if it was not associated with signs, symptoms, or treatment consistent with current guidelines [American Diabetes Association (ADA) 2005]. Severe hypoglycemia is defined as a hypoglycemic event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions (these episodes may be associated with sufficient neuroglycopenia to induce seizure or coma; also, BG measurements may not be available during such an event). Nocturnal hypoglycemia is defined as any hypoglycemic event that occurs between bedtime and waking.
Time Frame: Baseline through 24 weeks (wk) and 52 weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: events
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 268 | 267
events
  Total Events with BG ≤70 mg/dL,if available-24 wk | 10411 | 10976
  Total Events with BG ≤70 mg/dL,if available-52-wk | 19541 | 20852
  Severe Events-24 wk | 6 | 10
  Severe Events-52 wk | 13 | 16
  Nocturnal Events with BG ≤70 mg/dL-24 wk | 2217 | 2249
  Nocturnal Events with BG ≤70 mg/dL-52 wk | 4105 | 4485
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.703, Fisher Exact — P-value is for Total Events with BG ≤70 mg/dL,if available-24 wk
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.495, Fisher Exact — P-value is for Total Events with BG ≤70 mg/dL,if available-52-wk
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.174, Fisher Exact — P-value is for Severe Events-24 wk
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.828, Fisher Exact — P-value is for Severe Events-52 wk
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.661, Fisher Exact — P-value is for Nocturnal Events with BG ≤70 mg/dL-24 wk
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.606, Fisher Exact — P-value is for Nocturnal Events with BG ≤70 mg/dL-52 wk

13. Secondary Outcome: Rate Per 30 Days of Hypoglycemic Events
Description: The rate of hypoglycemic events per 30 days is defined as the total number of events between visits divided by the actual number of days between visits, and then multiplied by 30 days. A hypoglycemic event is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia, or has blood glucose (BG) concentration of ≤ 70 milligrams/deciliter [mg/dL (3.9 millimoles/liter (mmol/L)], even if it was not associated with signs, symptoms, or treatment consistent with current guidelines (ADA 2005). Severe hypoglycemia is defined as a hypoglycemic event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions (these episodes may be associated with sufficient neuroglycopenia to induce seizure or coma; also, BG measurements may not be available during such an event). Nocturnal hypoglycemia is defined as any hypoglycemic event that occurs between bedtime and waking.
Time Frame: Baseline through 24 weeks (wk) and 52 weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: hypoglycemic events per 30 days
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Number analyzed (Participants) | 268 | 267
hypoglycemic events per 30 days
  Total Events with BG ≤70 mg/dL, if available-24 wk | 7.10 (6.35) | 7.32 (6.58)
  Severe Events-24 wk | 0.00 (0.04) | 0.01 (0.04)
  Nocturnal Events with BG ≤70 mg/dL-24 wk | 1.50 (1.93) | 1.51 (1.77)
  Total Events with BG ≤70 mg/dL, if available-52 wk | 6.33 (5.64) | 6.56 (6.12)
  Severe Events-52 wk | 0.01 (0.04) | 0.01 (0.04)
  Nocturnal Events with BG ≤70 mg/dL-52 wk | 1.32 (1.66) | 1.42 (1.60)
Statistical Analysis 1: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.717, Wilcoxon (Mann-Whitney) — P-value is for Total Events with BG ≤70 mg/dL, if available-24 wk
Statistical Analysis 2: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.163, Wilcoxon (Mann-Whitney) — P-value is for Severe Events-24 wk
Statistical Analysis 3: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.669, Wilcoxon (Mann-Whitney) — P-value is for Nocturnal Events with BG ≤70 mg/dL-24 wk
Statistical Analysis 4: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.738, Wilcoxon (Mann-Whitney) — P-value is for Total Events with BG ≤70 mg/dL, if available-52 wk
Statistical Analysis 5: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.826, Wilcoxon (Mann-Whitney) — P-value is for Severe Events-52 wk
Statistical Analysis 6: Comparison: LY2963016 + Insulin Lispro vs Lantus + Insulin Lispro; Test type: Superiority or Other; p = 0.250, Wilcoxon (Mann-Whitney) — P-value is for Nocturnal Events with BG ≤70 mg/dL-52 wk

ADVERSE EVENTS:
Arm/Group | LY2963016 + Insulin Lispro | Lantus + Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 20/268 | 24/267
Other Adverse Events (participants affected / at risk) | 161/268 | 158/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2963016 + Insulin Lispro (N=268) | Lantus + Insulin Lispro (N=267)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) — Event resulted in death
Chest pain (General disorders) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 13 (16) | 12 (17)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gliomatosis cerebri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2963016 + Insulin Lispro (N=268) | Lantus + Insulin Lispro (N=267)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 12 (13) | 10 (16)
Gastritis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Toothache (Gastrointestinal disorders) | 4 (5) | 1 (3)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)
Fatigue (General disorders) | 4 (4) | 3 (4)
Influenza like illness (General disorders) | 3 (4) | 5 (6)
Injection site reaction (General disorders) | 3 (17) | 2 (3)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4) | 8 (9)
Cystitis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 8 (8) | 7 (7)
Gastroenteritis viral (Infections and infestations) | 5 (6) | 3 (3)
Influenza (Infections and infestations) | 5 (7) | 9 (9)
Nasopharyngitis (Infections and infestations) | 43 (68) | 45 (58)
Pharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Sinusitis (Infections and infestations) | 7 (8) | 8 (11)
Tooth abscess (Infections and infestations) | 1 (1) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 22 (24) | 21 (28)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 9 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Dizziness (Nervous system disorders) | 6 (7) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 7 (17)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (7)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
Hypertension (Vascular disorders) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days